CLINICAL TRIAL: NCT04849494
Title: Respiratory Morbidity of Late-Preterm Vs Intrauterine Growth Retarded Infants at School Age
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: TUTF-GOKAEK 2013/150.
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Intrauterine Growth Restriction; Preterm Birth
Keywords: Premature Birth; Late preterm; Fetal Growth Retardation; Asthma; School-age
MeSH Terms: conditions — Fetal Growth Retardation; Premature Birth; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Late preterm AGA infants/Group 1: According to the new BALLARD scoring system gestational age was 34-36 6/7 and those who were at the 10-90th percentile according to the Fenton growth curves
  Interventions: Other: ATS-DLD-78-C and ISAAC questionnaires
- Newborns with Intrauterine growth restriction/Group 2: Term or preterm infants below 10th percentile according to the values calculated according to Fenton growth curves
  Interventions: Other: ATS-DLD-78-C and ISAAC questionnaires
- Control/Group 3: the healthy term (gestation week 38-42 weeks), AGA newborns, who born between January 2006 and December 2008
  Interventions: Other: ATS-DLD-78-C and ISAAC questionnaires

INTERVENTIONS:
Other: ATS-DLD-78-C and ISAAC questionnaires — Early, natal and postnatal period data were recorded from the hospital database system and patient file. The morbidities observed during the follow-up of the newborns, the duration of hospitalization, needed of oxygen, surfactant administration, positive pressure ventilation requirement, and need for mechanical ventilation support and duration were noted from patient file records. Anthropometric measurements of all patients were taken. Demographic information, socioeconomic level, mother/father education level, mother's smoking status and medical history were questioned, and physical examinations of the patients were performed. were performed for screening respiratory diseases. After the physical examination, the validated Turkish forms of ATS-DLD-78-C and ISAAC questionnaires were filled in face-to-face by the research doctor who did not know the patients' medical history

SUMMARY:
Background: It is increasingly recognized that late preterm infants have increased respiratory morbidity in the neonatal period as well as decreased lung function in later life. Also, in-utero growth retardation (IUGR) and low birth weight are associated with increased respiratory morbidity beginning from infancy, throughout childhood and into adulthood. However, very few studies have assessed long term respiratory consequences of late preterm birth in comparison with IUGR.

Aim: To determine respiratory morbidity of late-preterm vs infants with IUGR at school age Study Design: Participants included late-preterm AGA infants (34-36, 6/7 weeks), IUGR infants (term/preterm) and term AGA infants born between 2004 and 2008 were included in this study and assessed for respiratory morbidity at school age. To assess the impact of late-preterm birth compared with IUGR and term gestation on respiratory morbidity by using a validated questionnaire. Wheezing, infectious respiratory morbidity and physician-diagnosed asthma panels were evaluated.

DETAILED DESCRIPTION:
Our study is a cross-sectional study in which the school-age respiratory morbidity of newborns with late preterm and IUGR birth history who were followed and treated by Trakya University Faculty of Medicine, Department of Pediatrics, Division of Neonatology between January 2006 and December 2008 were evaluated.

A total number of 160 children were included in the study. Children who admitted to the Neonatal intensive care unit and/or those who were born at the obstetrics unit and followed up with their mothers between January 2006 - December 2008 and reevaluated at school age (5-7 years old) during the study, were divided into two main groups: Late preterm AGA infants: according to the new BALLARD scoring system (5) gestational age was 34-36 6/7 and those who were at the 10-90th percentile according to the Fenton growth curves (6) (Group 1). Newborns with IUGR: term or preterm infants below 10th percentile according to the values calculated according to Fenton growth curves (6) (Group 2). In addition to these groups, preterm IUGR infants (<32 weeks of gestation) (Group 2a), and an equal number of preterm AGA infants (<32 weeks of gestation) (Group 3), late preterm (between 34-36 6/7 gestational weeks) IUGR infants (Group 2b) were divided into subgroups. And, the healthy term (gestation week 38-42 weeks), AGA newborns, who born between January 2006 and December 2008, were included in the study as a control group (Group 4) (Figure 1). The presence of major anomalies, patients who did not come to the school-age assessment or and rejected the informed consent form were excluded from the study.

Early (perinatal-neonatal), natal and postnatal period data were recorded from the hospital database system and patient file. The morbidities observed during the follow-up of the newborns, the duration of hospitalization, needed of oxygen, surfactant administration, positive pressure ventilation requirement, and need for mechanical ventilation support and duration were noted from patient file records. During the study, the study and control group cases who were at school age and had perinatal parameters as defined above were contacted by phone and invited to the outpatient clinic. Anthropometric measurements of all patients were taken (Tartımsan brand, TBS model, scale with serial number 1212430 and height meter). Demographic information, socioeconomic level, mother/father education level, mother's smoking status and medical history were questioned, and physical examinations of the patients were performed. The validated Turkish forms of ATS-DLD-78-C (7) and ISAAC questionnaires (8) were tested on 10 randomly selected patients by 2 different investigators to evaluate their intelligibility for screening respiratory diseases. The questionnaires were applied separately to both mother and father and after comparing the answers, it was decided that the questions were understandable. After the physical examination, the questionnaire forms were filled in face-to-face by the research doctor who did not know the patients' medical history (M.C.U).

Responses to the survey questions include; the presence of wheezing/wheezing in the chest independent of having a cold, presence of wheezing in the chest day/night, presence of two or more wheezing episodes causing shortness of breath, the need of using medication during wheezing attacks causing shortness of breath, one or more of the presence of wheezing episodes after exercise or playing games "Respiratory morbidity 1 included wheezing panel", presence of hospitalization due to severe respiratory infection under 2 years of age, having had more than 1 previous bronchiolitis/bronchitis/pneumonia or two or three of them, more than 3 days in the last 3 years of chest disease, cough/sputum attacks lasting at least for a week or longer, sputum, breast fullness, cough present for more than 3 months of the year "Respiratory morbidity 2 included previous infectious respiratory morbidity panel", presence of physician -diagnosed asthma history, current asthma, and the presence of a history of being followed up with a diagnosis of asthma "Respiratory morbidity 3 physician -diagnosed asthma panel" (9-13).

ELIGIBILITY:
Inclusion Criteria:

Children who admitted to the Neonatal intensive care unit and/or those who were born at the obstetrics unit and followed up with their mothers between January 2006 - December 2008 and reevaluated at school age (5-7 years old) during the study.

* None of major anomalies,
* Patients who come to the school-age assessment
* Accept the informed consent form

Exclusion Criteria:

* The presence of major anomalies,
* Patients who did not come to the school-age assessment
* Rejected the informed consent form

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total number of 160 children were included in the study. Children who admitted to the Neonatal intensive care unit and/or those who were born at the obstetrics unit and followed up with their mothers between January 2006 - December 2008 and reevaluated at school age (5-7 years old) during the study, were divided into two main groups: Late preterm AGA infants: according to the new BALLARD scoring system gestational age was 34-36 6/7 and those who were at the 10-90th percentile according to the Fenton growth curves. Newborns with IUGR: term or preterm infants below 10th percentile according to the values calculated according to Fenton growth curves. And, the healthy term (gestation week 38-42 weeks), AGA newborns, who born between January 2006 and December 2008, were included in the study as a control group
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2014-03-30 (Actual)

PRIMARY OUTCOMES:
to evaluate respiratory morbidity of late preterm and IUGR newborns at school age | between 5 to 7 years of age

SECONDARY OUTCOMES:
to point out the effects of risk factors encountered in the neonatal period for respiratory morbidity at school age | between 5 to 7 years of age

IPD SHARING:
Plan to Share IPD: Undecided
If there is an acceptable reason, Individual participant data (IPD) may be made available to other researchers, with the consent of patients.